CLINICAL TRIAL: NCT04590534
Title: Evaluation of the Effect of Garcinia in Combination With Chromium on the Clinical Outcomes of Patients With Symptomatic Benign Prostatic Hypertrophy
Brief Title: Evaluation of the Effect of Garcinia in Combination With Chromium on the Clinical Outcomes of Patients With LUTS/BPH
Acronym: BPH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Waleed El-Shaer, MD, Principal Investigator, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IDIRB2017122601-105
Record Dates: First submitted 2020-10-05; First posted 2020-10-19 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- study Group A (Experimental): patients will receive one capsule of [garcinia 500 mg and chromium 281 mg] 3 times daily for 12 weeks.
  Interventions: Drug: Chromax
- Active control Group B (Active Comparator): patients will receive one capsule of Sidosin 8 mg once daily for 12 weeks
  Interventions: Drug: Sildosin Group
- Placebo Group C (Placebo Comparator): patients will receive placebo 3 times daily for 12 weeks
  Interventions: Other: Placebo Group

INTERVENTIONS:
Drug: Chromax — Treatment of BPH by Chromax for 3 Months
  Other Names: study Group
  Arms: study Group A
Drug: Sildosin Group — patients will receive one capsule of Sidosin 8 mg once daily for 12 weeks
  Other Names: Active control Group A
  Arms: Active control Group B
Other: Placebo Group — patients will receive placebo 3 times daily for 12 weeks
  Other Names: Placebo Comparator
  Arms: Placebo Group C

SUMMARY:
To evaluate efficacy and safety of garcinia extract + chromium combinations (Chromax) in symptomatic benign prostatic hypertrophy patients

DETAILED DESCRIPTION:
Benign prostatic hypertrophy (BPH) can be defined as a slowly progressive prostatic adenoma that cause bladder outlet obstruction. Risk factors for BPH can be classified into modifiable risk factor including genetic factors and age with prevalence of 50% to 60% for males in their 60's up to 80% to 90% of those who are over 70 years of age, and non-modifiable risk factors including sex steroid hormones, the metabolic syndrome, obesity, diabetes, physical activity, diet, and inflammation. The clinical presentation of BPH can be categorized into storage and voiding abnormalities. Symptoms include urinary frequency and urgency, nocturia and dysuria in addition to urinary hesitancy, dribbling and incomplete bladder voiding. Several hypotheses are postulated to explain the pathophysiology of BPH including the testosterone and dihydrotestosterone, age related tissue remodelling, prostatic inflammation and metabolic aberration as obesity, diabetes and dyslipidemia.

Oxidative stress has been reported to play a role the pathogenesis of BPH. Oxidative stress has been considered to be one of the mechanisms that trigger the chain of reactions involved in the development and progression of prostatic hyperplasia. This is especially true as the human prostate tissue is vulnerable to oxidative DNA damage due to more rapid cell turnover and fewer DNA repair enzymes. In a study conducted on prostate tissue, it was observed that oxidative stress and oxidative DNA damage are important in the pathogenesis of BPH. Higher oxidative stress markers in terms of Malondialdehyde levels was reported in BPH patients. Moreover, a systematic review revealed that prostatic inflammation can induce free radicals formation that might play role in carcinogenesis and development of prostate cancer in patients with BPH.

Garcinia cambogia is a natural fruit which has been reported to have anti-obesity activity including reduced food intake and body fat gain by regulating the serotonin levels related to satiety, increased fat oxidation and decreased de novo lipogenesis. It also exerted hypolipidemic, antidiabetic, anti-inflammatory, anticancer, anthelmintic, anticholinesterase and hepatoprotective activities in in vitro and in vivo models . Hydro-citric acid, the main component of garcinia extract, has been reported to have strong antioxidant property.

An animal study on rats has reported that kolaviron, a bioflavonoid complex from Garcinia kola had decreased prostate weights (compared with the normal control and reversed the histoarchitecture of the prostates of the BPH rats.

ELIGIBILITY:
Inclusion Criteria:

* LUTS/BPH

Exclusion Criteria:

* Previous prostatic surgery or radiation therapy.
* Treatment with anti-BPH drugs within a month before the beginning of study (washout) or, 5α-reductase inhibitor (5-ARI) use within 6 months prior to entry, use of drugs like LHRH.
* Patient receiving chromium and garcinia extract before inclusion in the study.
* complicated LUTS/BPH requring surgical treatment Neurogenic Bladder

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-03-12 (Estimated)

PRIMARY OUTCOMES:
1-International prostate symptoms score(IPSS) | change of baseline and 3 months post-treatment
  IPSS score Ranges from1 to 35, lower score is better

SECONDARY OUTCOMES:
2- Volume of prostate(PV) | change of PV from baseline and 3 months post-treatment
  2- measred prostate Volume mesured by transrectal ultra sound (normal 20+- 5)
4- Residual urine volume(PVRU) | Change of PVRU from baseline and 3 months post-treatment
  Post voiding Residual urine volume normally about 0
Prostativ Specific Antigen (PSA) | Change of PSA from baseline to 3 months post-treatment
  PSA normally up to 4.5 ng/ml
Body Mass index (BMI) | Change of BMI from baseline and 3 months post-treatment
  BMI is about 25

OTHER OUTCOMES:
Quality of life(QOL) | Change of QOL from baseline and 3 months post-treatment
  QOL Ranges 1 to 6 lower values is better

CONTACTS AND LOCATIONS:
Overall Officials: Waleed El-Shaer, M.D, Principal Investigator — Banha Univesity
Locations (1):
- Banha University Hospitals, Banhā, Kalubyia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Shaer W, Abd-Allah AR, El-Shafie MF, Salama IM, El Shaer A. Evaluation of the Therapeutic Potential of Garcinia cambogia Alone or in Combination With Silodosin in the Management of LUTS/BPH: A Prospective Randomized Controlled Study. Urology. 2025 Jun;200:198-205. doi: 10.1016/j.urology.2025.04.012. Epub 2025 Apr 8. PMID 40209997